CLINICAL TRIAL: NCT06186232
Title: Evaluation Of Bone Regenerated After Guided Bone Regenration (GBR) Using Customized 3D Printed Polymethylmethacrylate (PMMA) Membrane in Horizontally Deficient Maxillary Aesthetic Zone
Brief Title: Evaluation of Bone Regenerated With Guided Bone Regeneration (GBR) Using Polymethylmethacrylate (PMMA) Membrane
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Mohamed Sherif Abdel Mawgood, Evaluation Of Bone Regenerated After Guided Bone Regenration (GBR) using customized 3D printed Polymethylmethacrylate (PMMA) membrane in horizontally deficient maxillary aesthetic zone., Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS 3310
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Horizontal Ridge Deficiency
Keywords: polymethylmethacrylate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with horizontally deficient ridge in ethetic maxilary zone need (GBR) and implant placement (Other): a group of patients with with horizontally deficient ridge in esthetic maxillary zone will undergo ridge augmentation with guided bone regeneration (GBR) technique using polymethylmethacrylate (PMMA) polymer as membrane.
  Interventions: Procedure: guided bone regeneration (GBR).

INTERVENTIONS:
Procedure: guided bone regeneration (GBR). — guided bone regeneration (GBR) using polymethylmethacrylate (PMMA) polymer as membrane.
  Other Names: implant installation 6 months after (GBR)

SUMMARY:
To evaluate the quantity and quality of bone generated, radiographically and histomorphometrically, after guided bone regeneration (GBR) using a membrane of 3D printed custom made (PMMA) and subsequent stability of delayed implant placement.

DETAILED DESCRIPTION:
Guided bone regeneration (GBR), is the most widely used technique to facilitate bone generation. It depends on using a biocompatible membrane that acts as physical barrier preventing the connective tissue from invading the bone defect.

To achieve maximum bone regeneration, GBR membrane should have several characteristics, including:

* Biocompatibility.
* Proper stiffness for space maintenance.
* Prevent epithelial cell migration.
* Appropriate resorption time after proper bone regeneration. Membranes used in guided bone regeneration (GBR) may have some limitations as the need of second surgery for removal of the membrane (in case of non-resorbable membranes as titanium mesh or expanded polytetrafluoroethylene (e-PTFE) membranes), lake of space maintenance (as collagen membranes) in addition to their high cost.

Thus, we aim to use a commercially available material as polymethyl methacrylate (PMMA) with (GBR) to facilitate bone generation as well as subsequent implant placement.

Recent forms of (PMMA), have been certified to be biocompatible and safe for skin and mucosal contact. PMMA is characterized by having high toughness which may provide a space maintenance when using as membrane in guided bone regeneration (GBR). The PMMA prosthesis can be pre-fabricated, which results in reduction of surgical time, easy technical handling and good esthetic results.

In addition, it has a relatively low cost when it is compared to other types of membranes used in guided bone regeneration (GBR).

ELIGIBILITY:
Inclusion Criteria:

* Patients with edentulous area related to horizontally deficient aesthetic zone of maxilla.
* Patients are physically healthy with no medical history of any systemic or local disease that would contraindicate ridge augmentation and/or implant surgery or complicate the healing process. (Severe liver or kidney disease, a history of head and neck radiotherapy, chemotherapy at the time of surgery, uncontrolled diabetes, active periodontal in the residual dentition, inflammatory or autoimmune disorders of the oral mucosa, poor oral hygiene, patient failure to cooperate, and any other disease condition contraindicating the oral surgery).
* Non-smokers.
* Free from temporomandibular joint disorders and abnormal oral habits such as bruxism.
* The edentulous ridges were covered with optimal thickness of keratinized mucosa with no signs of inflammation, ulceration or scar tissue.
* The occlusion shows sufficient inter-arch space for future prothesis.

Exclusion Criteria:

* General contraindications to surgery.
* Patients subjected to irradiation in the head and neck area less than 1 year before fixation.
* Untreated periodontitis.
* Poor oral hygiene.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Patients participating in other studies, if the present protocol could not be properly followed

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
amount of bone gain | 6 months postoperative
  radiographic using cone beam computed tomography (CBCT)

SECONDARY OUTCOMES:
quality of bone regenerated | 6 months after surgical procedure
  bone core biopsy (histomorphometric analysis)

OTHER OUTCOMES:
post operative ridge width | 6 months postoperative
  using bone caliper
initial implant stability | 6 months post operative
  using manual ratchet

CONTACTS AND LOCATIONS:
Overall Officials: Hesham El Hawary, Study Director — Professor of Oral and Maxillofacial surgery, Cairo university

REFERENCES:
- [Background] Khojasteh A, Kheiri L, Motamedian SR, Khoshkam V. Guided Bone Regeneration for the Reconstruction of Alveolar Bone Defects. Ann Maxillofac Surg. 2017 Jul-Dec;7(2):263-277. doi: 10.4103/ams.ams_76_17. PMID 29264297
- [Background] Benic GI, Hammerle CH. Horizontal bone augmentation by means of guided bone regeneration. Periodontol 2000. 2014 Oct;66(1):13-40. doi: 10.1111/prd.12039. PMID 25123759
- [Background] Elgali I, Omar O, Dahlin C, Thomsen P. Guided bone regeneration: materials and biological mechanisms revisited. Eur J Oral Sci. 2017 Oct;125(5):315-337. doi: 10.1111/eos.12364. Epub 2017 Aug 19. PMID 28833567
- [Background] Lee SW, Kim SG. Membranes for the Guided Bone Regeneration. Maxillofac Plast Reconstr Surg. 2014 Nov;36(6):239-46. doi: 10.14402/jkamprs.2014.36.6.239. Epub 2014 Nov 12. PMID 27489841
- [Background] Fernandes da Silva AL, Borba AM, Simao NR, Pedro FL, Borges AH, Miloro M. Customized polymethyl methacrylate implants for the reconstruction of craniofacial osseous defects. Case Rep Surg. 2014;2014:358569. doi: 10.1155/2014/358569. Epub 2014 Jun 30. PMID 25093139
- [Background] Freitas de Andrade P, Meza-Mauricio J, Kern R, Faveri M. Labial Repositioning Using Print Manufactured Polymethylmethacrylate- (PMMA-) Based Cement for Gummy Smile. Case Rep Dent. 2021 Dec 21;2021:7607522. doi: 10.1155/2021/7607522. eCollection 2021. PMID 34970460
- [Background] AlSubaie MF, Al-Sharydah AM, Nassim HM, Alhawsawi A. Orbital Floor Blowout Fracture Reconstruction Using Moldable Polymethyl Methacrylate: A Report of Two Cases and Their Imaging Findings. Open Access Emerg Med. 2022 May 25;14:223-232. doi: 10.2147/OAEM.S359173. eCollection 2022. PMID 35656329